CLINICAL TRIAL: NCT04255628
Title: The Brain Metabolic Change in Chronic Cancer Pain Patient: FDG PET Image Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201911071RINC
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-01

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with cancer pain: head and neck and esophageal cancer patients. with cancer pain
  Interventions: Diagnostic Test: FDG PET
- without cancer pain: head and neck and esophageal cancer patients. without cancer pain=30
  Interventions: Diagnostic Test: FDG PET

INTERVENTIONS:
Diagnostic Test: FDG PET — Cancer patients who scheduled whole body FDG-PET image scan for clinically indicated.

SUMMARY:
Cancer pain deteriorated in quality of life and related with numerous psychosocial problems. Over the one third of cancer patient suffered from moderate to severe cancer pain, even under adequate pain management.

The 18F-fluoro-2-deoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) images can provide quantitative results in clinical oncology. As a functional neuroimaging, the PET evidently provided anatomical activated regions, size, and spatial extent information. In this study, we use FDG-PET to investigate changes concerning the glucose metabolism in the brain with or without cancer pain. Therefore, we may provide useful information to treatment target in cancer pain patients.

DETAILED DESCRIPTION:
Overall, cancer incidence has decreased and the rate of cancer deaths in both men and women has also significantly declined among both men and women in all site.However, the prevalence of chronic pain is 28.2%, ranging from 22.5% to 35.4%, depending on the location of the primary tumor, and neuropathic characteristics were observed in 19.9% of patients with chronic cancer pain.

Despite numerous studies on cancer pathogenesis and diagnosis, few reports have demonstrated the brain mechanism underlying cancer pain. One study used resting functional magnetic resonance imaging (fMRI) to identify the changes in the functional brain network of chronic bone cancer pain mice under anesthesia. Cancer-induced bone pain (CIBP) might alter resting state activity of the cingulate cortex, prefrontal cortex (PFC) and ventral striatum, indicating a strong affective component of the CIBP mice.In imaging studies of human patients with cancer, patients with chronic cancer pain exhibited activation in the PFC.

The 18F-fluoro-2-deoxyglucose (FDG) positron emission tomography/computed tomography (PET/CT) images can provide quantitative results in clinical oncology.Owing to the higher glucose metabolic rate in the brain, brain FDG-PET images are not routinely used in the clinical setting. However, several studies have demonstrated functional brain changes in human pain condition.In this study, we use FDG-PET to investigate changes concerning the glucose metabolism in the brain with or without cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients who scheduled whole body FDG-PET image scan for clinically indicated.
2. Age > 20

Exclusion Criteria:

1. Unable to complete questionnaires.
2. Prior evidence of brain metastases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients in each group of head and neck and esophageal cancer patients. Each cancer group include without cancer pain=30, with cancer pain=30.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
Brain metabolism change | 12 months
  The FDG-PET of Standardized uptake values (SUVs) were calculated for each voxel in the reconstructed images to investigate changes concerning the glucose metabolism in the brain with or without cancer pain

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hosipital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol